CLINICAL TRIAL: NCT05751408
Title: Technical Evaluation of Commercial IMUs Within Clinical Gait Analysis in Adult Patients With Neurological Disorders
Brief Title: Technical Evaluation of Commercial IMUs Within Clinical Gait Analysis
Status: Recruiting | Type: Observational
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-16038
Record Dates: First submitted 2023-01-25; First posted 2023-03-02 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Gait Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stiff knee gait: Subjects referred to clinical 3D gait analysis because of a clinical question related to stiff knee gait
  Interventions: Procedure: gait analysis using 3D (Vicon) and IMU (Movella)
- Foot surgery: Subjects referred to clinical 3D gait analysis because of a clinical question related to foot surgery
  Interventions: Procedure: gait analysis using 3D (Vicon) and IMU (Movella)

INTERVENTIONS:
Procedure: gait analysis using 3D (Vicon) and IMU (Movella) — Subjects are measured using Vicon 3D analysis, combined with IMU-sensors

SUMMARY:
A standard clinical gait analysis consists of observing walking with video (2D) or advanced equipment (VICON 3D). This 3D method provides detailed information about the gait pattern, but is time-consuming in implementation and data analysis. There are commercial 3D systems on the market that are used in healthy individuals and in sports. These so-called Inertial Measurement Units (IMUs) may also be suitable for use in the clinic. In this research protocol, the aim is to test the usability of commercial sensors and technically compare them with standard clinical 3D gait analysis in adult patients with a neurological disorder.

DETAILED DESCRIPTION:
Measurements will include subjects that perform routine clinical 3D gait analysis because of a clinical question related to stiff knee gait or surgical intervention of the foot. During routine clinical gait analysis, Vicon markers and EMG-measurements of specified muscles is included. IMU-sensors will be included to this routine measurements to measure accelorometer, gyroscope and magnetometer data of both feet, both upper and lower legs, the sternum and the sacrum.

ELIGIBILITY:
Subjects referred for clinical gait analysis at Roessingh Centre for Rehabilition in Enschede, the Netherlands:

Inclusion Criteria:

* Disorders affecting walking, including amongst others stroke, traumatic brain injury, MS, incomplete spinal cord injury, CP, Spina Bifida, neuromuscular diseases
* age minimum 18 years
* Viosca score minimum 2; meaning minimal independent walking ability indoors
* increased fall risk or increased effort of walking because of: 1) decreased stability during stance; and/or 2) decreased foot clearance during swing; and/or 3) not able to walk on bare feet because of equinovarus; and/or 4) fatigue during walking because of compansatory strategies.

Exclusion Criteria:

* subjects referred for clinical gait analysis because of problems other than stiff knee gait or foot surgery
* severe deficits in communication, memory and understanding at such a level that it would affect instructions during the measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects minimum 18 years of age, referred for clinical gait analysis at Roessingh, Centre for Rehabilitation in Enschede, the Netherlands with disorders affecting walking, including amongst others stroke, traumatic brain injury, MS, incomplete spinal cord injury, CP, Spina Bifida, neuromuscular diseases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Ankle angle assessed by Vicon | baseline
  Vicon 3D analysis will be used to assess ankle angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Ankle angle assessed by Vicon | 1 year
  Vicon 3D analysis will be used to assess ankle angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Knee angle assessed by Vicon | baseline
  Vicon 3D analysis will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Knee angle assessed by Vicon | 1 year
  Vicon 3D analysis will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Hip angle assessed by Vicon | baseline
  Vicon 3D analysis will be used to assess hip angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Hip angle assessed by Vicon | 1 year
  Vicon 3D analysis will be used to assess hip angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Ankle angle assessed by IMU sensors | baseline
  IMU sensors will be used to assess ankle angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Ankle angle assessed by IMU sensors | 1 year
  IMU sensors will be used to assess ankle angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Knee angle assessed by IMU sensors | baseline
  IMU sensors will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Knee angle assessed by IMU sensors | 1 year
  IMU sensors will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Hip angle assessed by IMU sensors | baseline
  IMU sensors will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)
Hip angle assessed by IMU sensors | 1 year
  IMU sensors will be used to assess knee angles (in degrees) during walking. Angles will be defined from the moment the foot hits the ground (initial contact) until the foot hits the ground again (second initial contact)

SECONDARY OUTCOMES:
Age | at inclusion
  Age (in years)
Height | at inclusion
  Height (in cm)
Weight | at inclusion
  Weight (in kg)
FAC-score | at inclusion
  Functional Ambulation Categorie score (0-5 points) to assess independence of walking

CONTACTS AND LOCATIONS:
Overall Officials: C Nikamp, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: No